CLINICAL TRIAL: NCT03896763
Title: PROSpect: Prone and Oscillation Pediatric Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University Medical Center Groningen (Other); Boston Children's Hospital (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Martha A.Q. Curley, PhD, RN, Ruth M. Colket Endowed Chair in Pediatric Nursing, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 831295; 5UH3HL141736-03 (NIH)
Record Dates: First submitted 2018-10-22; First posted 2019-04-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Acute Respiratory Distress Syndrome in Children
Keywords: Pediatric Acute Respiratory Distress Syndrome (PARDS); Acute Respiratory Distress Syndrome (ARDS); acute respiratory failure; child; pediatric intensive care unit
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: Two-by-two factorial, response-adaptive, randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supine / CMV (Experimental): Supine positioning and conventional mechanical ventilation
  Interventions: Other: Either supine or prone positioning and either CMV or HFOV
- Prone / CMV (Experimental): Prone positioning and conventional mechanical ventilation
  Interventions: Other: Either supine or prone positioning and either CMV or HFOV
- Supine / HVOF (Experimental): Supine positioning and high-frequency oscillatory ventilation
  Interventions: Other: Either supine or prone positioning and either CMV or HFOV
- Prone / HFOV (Experimental): Prone positioning and high-frequency oscillatory ventilation
  Interventions: Other: Either supine or prone positioning and either CMV or HFOV

INTERVENTIONS:
Other: Either supine or prone positioning and either CMV or HFOV — Supine positioning: Subjects randomized to supine positioning will remain supine.
  Prone positioning: Subjects randomized to prone positioning will be positioned prone ≥16 hours/day for a maximum of 28 days.
  CMV strategy: Low tidal volume to obtain exhaled Vt of 5-7 ml/kg (ideal body weight), PIP goal limited to ≤ 28 cm H2O and lung recruitment maneuver to identify best PEEP then maintained per PEEP-FiO2 grid.
  HFOV strategy: Frequency at 8-12 Hz, amplitude (delta-P) 60-90 and mPaw recruitment maneuver.
  Other Names: Supine positioning; Prone positioing; Conventional mechanical ventilation (CMV); High frequency oscillatory ventilation (HFOV)

SUMMARY:
Severe pediatric acute respiratory distress syndrome (PARDS) is a life-threatening and frequent problem experienced by thousands of children each year. Little evidence supports current supportive practices during their critical illness. The overall objective of this study is to identify the best positional and/or ventilation practice that leads to improved patient outcomes in these critically ill children. We hypothesize that children with high moderate-severe PARDS treated with either prone positioning or high-frequency oscillatory ventilation (HFOV) will demonstrate more days off the ventilator when compared to children treated with supine positioning or conventional mechanical ventilation (CMV).

DETAILED DESCRIPTION:
PROSpect is a two-by-two factorial, response-adaptive, randomized controlled clinical trial of supine/prone positioning and conventional mechanical ventilation (CMV)/high-frequency oscillatory ventilation (HFOV). About 60 pediatric intensive care units (PICUs), two thirds U.S. and one third international, with at least 5 years of experience with prone positioning and HFOV in the care of pediatric patients with severe Pediatric Acute Respiratory Distress Syndrome (PARDS), that can provide back-up extracorporeal membrane oxygenation (ECMO) support, are participating. Eligible consecutive subjects with high moderate-severe PARDS will be randomized to one of four groups: supine/CMV, prone/CMV, supine/HFOV, prone/HFOV. Subjects who fail their assigned positional and/or ventilation therapy for either persistent hypoxia or hypercapnia may receive the reciprocal therapy while being considered for ECMO cannulation. Our primary outcome is ventilator-free days (VFD) through day 28, where non-survivors receive zero VFD. We hypothesize that children with severe PARDS treated with either prone positioning or HFOV will demonstrate ≥ 2 more VFD. Our secondary outcome is nonpulmonary organ failure-free days. We will also explore the interaction effects of prone positioning with HFOV on VFDs and also investigate the impact of these interventions on 90-day in-hospital mortality and, among survivors, the duration of mechanical ventilation, PICU and hospital length of stay, and the trajectory of post-PICU functional status and health-related quality of life (HRQL). Up to 600 subjects with severe PARDS will be randomized, stratified by age group and direct/indirect lung injury. Adaptive randomization will first occur after 300 patients are randomized and have been followed for 28 days, and every 100 patients thereafter. At these randomization update analyses, new allocation probabilities will be computed based on ongoing intention-to-treat trial results, increasing allocation to well performing arms and decreasing allocation to poorly performing arms. Data will be analyzed per intention-to-treat for the primary analyses and per-protocol received for primary, secondary and exploratory analyses.

ELIGIBILITY:
Inclusion criteria:

Intubated and mechanically ventilated with high moderate-severe PARDS for <48 hours per PALICC guidelines (chest imaging consistent with acute pulmonary parenchymal disease and OI ≥12 or OSI ≥10). We require two blood gases meeting moderate-severe PARDS criteria (separated by at least 4 ± 2 hours during which time the clinical team is actively working to recruit lung volume and optimize the patient's hemodynamic status per PALICC guidelines; specifically, incremental and decremental PEEP changes to optimize lung volume). A second blood gas is not required for OI ≥16.

Exclusion criteria:

* Perinatal related lung disease
* Unrepaired congenital diaphragmatic hernia or congenital/acquired diaphragm paralysis
* Respiratory failure explained by cardiac failure or fluid overload
* Cyanotic heart disease
* Cardiomyopathy
* Unilateral lung disease
* Primary pulmonary hypertension
* Intubated for status asthmaticus
* Obstructive airway disease (e.g., Severe airways disease without parenchymal involvement or disease characterized by hypercapnia with FiO2 <0.30 and/or evidence of increased resistance visible on the flow - time scalar and/or presence of intrinsic PEEP)
* Active air leak
* Bronchiolitis obliterans
* Post hematopoietic stem cell transplant; specifically, patients receiving continuous supplemental oxygen for three or more days prior to intubation; receiving noninvasive ventilation for more than 24 hours prior to intubation; receiving more than one vasoactive medication at time of meeting inclusion criteria; spending more than four days in the PICU prior to intubation; supported on or with immediate plans for renal replacement therapies; with two or more allogeneic transplants; who relapsed after the transplant; or with diffuse alveolar hemorrhage
* Post lung transplant
* Home ventilator dependent with baseline Oxygen Saturation Index (OSI) >6
* Neuromuscular respiratory failure
* Critical airway (e.g., post laryngotracheal surgery or new tracheostomy) or anatomical obstruction of the lower airway (e.g., mediastinal mass)
* Facial surgery or trauma in previous 2 weeks
* Head trauma (managed with hyperventilation)
* Intracranial bleeding
* Unstable spine, femur or pelvic fractures
* Open abdomen
* Currently receiving more than 6 consecutive hours of either prone positioning or HFOV
* Supported on ECMO during the current admission
* Family/medical team not providing full support (patient treatment considered futile)
* Previously enrolled in current study
* Enrolled in any other interventional clinical trial not approved for co-enrollment
* Known pregnancy

Ages: 2 Weeks to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Ventilator-free Days (VFD) | 28 days
  Our primary research hypothesis is that children with severe PARDS randomized to either prone positioning or HFOV will demonstrate more ventilator-free days. We hypothesize that a superior treatment would improve VFD by at least 2 days, a clinically meaningful difference. VFD is the number of days within 28 days that a patient is alive and free of mechanical ventilation. Improvement in VFD will be considered within the context of patient safety; specifically, patients must also exhibit a similar safety profile.

SECONDARY OUTCOMES:
Nonpulmonary organ failure-free days (OFFD) | 28 days
  Our secondary research hypothesis is that children with severe PARDS randomized to either prone positioning or HFOV will demonstrate more more nonpulmonary organ failure-free days. OFFD is the number of days within 28 days that a patient is alive and free of clinically significant non-pulmonary organ failure. Nonpulmonary organ failure-free days will be calculated based on the clinically important nonpulmonary organ systems (neurologic, cardiovascular, renal and hematologic) using nonpulmonary PEdiatric Logistic Organ Dysfunction-2 (PELOD-20 scores.

OTHER OUTCOMES:
Interaction effects of prone positioning with HFOV on VFDs - number of ventilator-free days | 28 days
  The number of ventilator-free days (VFD) will be compared between children randomized to prone/CMV and supine/HFOV to those randomized to prone/HFOV. VFD is the number of days within 28 days that a patient is alive and free of mechanical ventilation.
90-day in-hospital mortality | 90 days
  Deaths from all causes will be monitored through hospital discharge or day 90 (whichever occurs first). The primary and secondary causes of death (as specified on the death certificate) will be recorded to allow us to probe the cause of death in PARDS.
Duration of mechanical ventilation (among survivors) | 28 days, 90 days
  Duration of mechanical ventilation provides a prospective evaluation of ventilator support independent of mortality. The duration of mechanical ventilation is defined as the time from day 0 (intubation) to the first time the endotracheal tube is continuously absent for at least 24 hours. For subjects with tracheostomies, duration of mechanical ventilation is defined as the time of initiation of assisted breathing to the first time positive pressure is <5 cm H2O (continuous or bi-level) for at least 24 hours. Duration of mechanical ventilation will be considered to be 28 days for subjects still intubated on day 28, and will be calculated for subjects who survive to hospital discharge or day 90 (whichever occurs first).
PICU and hospital length of stay (among survivors) | 90 days
  PICU length of stay (LOS) is defined as the time from day 0 (intubation) to the time of PICU discharge, while hospital LOS is defined as the time from day 0 to the time of hospital discharge. PICU and hospital LOS will be considered to be 90 days for subjects still in the PICU/hospital on day 90, and will be calculated for subjects who survive to hospital discharge or day 90 (whichever occurs first).
Post PICU discharge functional status | 1, 3, 6, 12 months post PICU discharge
  Pre and post PICU functional status will be compared. Functional status will be assessed using the Pediatric Cerebral Performance (PCPC), Pediatric Overall Performance Category (POPC) and Functional Status Scale (FSS) score. The PCPC and POPC quantify short-term cognitive impairments and functional morbidity. Scores range from 1 to 6 for both scales with 1: good, 2: mild disability, and 6: brain death. The FSS is a valid and reliable assessment method to quantify functional status. The FSS includes 6 domains: mental status, sensory functioning, communication, motor function, feeding, and respiratory. Scores for each domain range from 1 (normal) to 5 (very severe dysfunction) with total scores ranging from 6 to 30.
Post PICU discharge health-related quality of life (HRQL) | 1, 3, 6, 12 months post PICU discharge
  Pre and post PICU health-related quality of life will be compared using the PedsQL 4.0 Generic Core Scales and Infant Scales - Acute Version They are 23-item child self-report and parent proxy-report scales with four domains: physical functioning, emotional functioning, social functioning, and school functioning. Scale ranges from 0 to 100, with higher scores indicating fewer problems. The PedsQL Infant Scales consist of 36-45 questions, depending on age, with 5 domains: physical functioning, physical symptoms, emotional functioning, social functioning, and cognitive functioning. The PedsQL™ Multi-dimensional Fatigue Scale - Acute Version is an 18-item scale that encompasses three domains: General Fatigue, Sleep/Rest Fatigue and Cognitive Fatigue. Higher scores indicate better HRQOL. PedsQL Pediatric Pain Questionnaire is a generic pain instrument. Subjects capable of self-reporting identify a point on a 100 mm line that best shows the worst pain they experienced in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Martha AQ Curley, RN, PhD, Principal Investigator — University of Pennsylvania; Ira M. Cheifetz, MD, Principal Investigator — UH Rainbow Babies and Children's Hospital; Martin CJ Kneyber, MD, PhD, Principal Investigator — Beatrix Children's Hospital; David Wypij, PhD, Principal Investigator — Boston Children's Hospital
Locations (49):
- United States (28):
  - Children's of Alabama, Birmingham, Alabama
  - Banner Health, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Orange County, Orange, California
  - Stanford Children's Health, Palo Alto, California
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - University of Iowa Stead Family Chlldren's Hospital, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Bloomberg Children's Center, Johns Hopkins University, Baltimore, Maryland
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital and Medical Center, Omaha, Nebraska
  - Cohen Children's Medical Center, Queens, New York
  - Duke Children's Hospital, Durham, North Carolina
  - UH Rainbow Babies & Children, Cleveland, Ohio
  - Children's Hospital at Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Medical City Dallas, Dallas, Texas
  - Children's Health Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - American Family Children's Hospital, University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital de Pediatría J. P. Garrahan. SAMIC, Buenos Aires, Buenos Aires F.D., Argentina
- Australia (2):
  - Perth Children's Hospital, Perth, Western Australia
  - Children's Hospital at Westmead, Sydney
- Brazil (2):
  - Sabara Hospital Infantil, São Paulo, Brazil
  - Hospital SEPACO, São Paulo
- Centre Hospitalier Universitaire Sainte Justine, Montreal, Quebec, Canada
- Münster University Hospital, Münster, Germany
- Rainbow Children's Hospital, Hyderabad, India
- Hadassah Medical Center, Jerusalem, Israel
- Italy (3):
  - Meyer Children's Hospital, Florence, Italy
  - Bambino Gesu Children's Hospital (Area Rossa Unit), Rome, Italy
  - Instituto Giannina Gasilini, Genova
- University of Malaysia Medical Center, Kuala Lumpur, Malaysia
- University Medical Center Groningen, Groningen, Netherlands
- Chonnam National University Hospital, Gwangju, South Korea
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok
  - Faculty of Medicine Ramathibodi Hospital, Bangkok
- Shaikh Khalifa Medical City, Abu Dhabi, United Arab Emirates
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham, UK
  - University Hospital Leicester NHS Trust, Leicester

IPD SHARING:
Plan to Share IPD: Yes
Per NHLBI policy, we will provide a deidentified dataset and all the data-related documentation necessary to utilize the study data (dictionary, calculated variables and standard operating procedures) to the NHLBI. We will submit this dataset to the NHLBI Data Repository managed by the BioLINCC (Biologic Specimen and Data Repository Information Coordinating Center).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years after the final follow-up interview or 2 years after the primary paper has been published, whichever comes first.
Access Criteria: Subject to the approval of the (1) PROSpect Ancillary Study Committee, (2) PROSpect Executive Committee, and (3) National Heart, Lung, and Blood Institute (NHLBI).

REFERENCES:
- [Derived] Kneyber MCJ, Cheifetz IM, Asaro LA, Graves TL, Viele K, Natarajan A, Wypij D, Curley MAQ; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Protocol for the Prone and Oscillation Pediatric Clinical Trial ( PROSpect ). Pediatr Crit Care Med. 2024 Sep 1;25(9):e385-e396. doi: 10.1097/PCC.0000000000003541. Epub 2024 May 28. PMID 38801306
- See also: Study Website — http://www.prospect-network.org/

DOCUMENTS (3):
  • Study Protocol (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT03896763/Prot_007.pdf
  • Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT03896763/SAP_005.pdf
  • Informed Consent Form (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/63/NCT03896763/ICF_006.pdf